CLINICAL TRIAL: NCT00014664
Title: A Phase II, Open-Label, Randomized, Multicenter Trial To Evaluate The Preliminary Safety And Efficacy of Hu1D10 In Patients With Relapsed Or Refractory Grades I, II, or III B-Cell Non-Hodgkin's Lymphoma (Including Follicular, Small Lymphocytic And Marginal Zone/MALT)
Brief Title: Monoclonal Antibody Therapy in Treating Patients With Relapsed or Refractory Non-Hodgkin's Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: PDL BioPharma, Inc. (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000068585; PDL-1D10-901; CUMC-0101-552
Record Dates: First submitted 2001-04-10; First posted 2003-06-10 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2002-09

CONDITIONS: Lymphoma
Keywords: recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — apolizumab

INTERVENTIONS:
Biological: apolizumab

SUMMARY:
RATIONALE: Monoclonal antibodies can locate cancer cells and either kill them or deliver cancer-killing substances to them without harming normal cells.

PURPOSE: Randomized phase II trial to compare the effectiveness of two different monoclonal antibody regimens in treating patients who have relapsed or refractory non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the relative safety of 3 different regimens of monoclonal antibody Hu1D10 in patients with relapsed or refractory grade I, II, or III B-cell non-Hodgkin's lymphoma.
* Compare the preliminary tumor response and progression-free survival of patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are randomized to 1 of 3 treatment arms.

* Arm I: Patients receive monoclonal antibody (MOAB) Hu1D10 IV over approximately 2 hours on days 1, 8, 15, and 22.
* Arm II: Patients receive MOAB Hu1D10 as in arm I at a higher dose.
* Arm III:Patients receive MOAB Hu1D10 IV on days 1, 3, 5, 8, 10, 12, 15, 17, 19, 22, 24, and 26.

Treatment in all arms continues in the absence of disease progression or unacceptable toxicity.

Patients are followed at weeks 1, 4, and 12 and then at months 6, 9, 12, 18, and 24.

PROJECTED ACCRUAL: A total of 60 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed relapsed or refractory grade I, II, or III non-Hodgkin's lymphoma (NHL), including follicular, small lymphocytic, or marginal zone/MALT lymphoma
* Previously treated with radiotherapy, immunotherapy, and/or chemotherapy for NHL

  * Progression of disease or no response since last treatment for NHL
* 1D10+ lymphoma by immunohistochemistry or flow cytometry
* Bidimensionally measurable disease at least 2 cm in a single dimension
* No CNS metastases
* Circulating tumor cells no greater than 5,000/mm^3

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* At least 3 months

Hematopoietic:

* Platelet count at least 75,000/mm^3 (unless disease related)
* Neutrophil count at least 1,000/mm^3 (unless disease related)
* Hemoglobin greater than 8.0 g/dL

Hepatic:

* Bilirubin less than 2.5 mg/dL
* SGOT less than 4 times upper limit of normal

Renal:

* Creatinine less than 2.5 mg/dL

Cardiovascular:

* No clinically significant cardiac disease (New York Heart Association class III or IV)
* No evidence of myocardial infarction or cardiac arrhythmia (unless surgically repaired) within the past 6 months

Pulmonary:

* No clinically significant pulmonary disease

Other:

* No other malignancy within the past 2 years except non-melanoma skin cancer or carcinoma in situ
* No significant psychiatric or CNS impairment
* No active serious infection
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 1 month after study
* Negative anti-Hu1D10 antibody response (HAHA/HAMA)
* HIV negative

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Disease Characteristics
* At least 4 weeks since prior interferon therapy
* At least 3 months since prior immunotherapy
* No prior monoclonal antibody Hu1D10

Chemotherapy:

* See Disease Characteristics
* At least 4 weeks since prior cytotoxic chemotherapy

Endocrine therapy:

* At least 4 weeks since prior corticosteroids (more than 10 mg prednisone/day)
* No concurrent corticosteroids at more than 10 mg prednisone/day for pre-existing diseases or adverse reactions

Radiotherapy:

* See Disease Characteristics
* At least 4 weeks since prior external beam radiotherapy
* At least 3 months since prior radioimmunotherapy

Surgery:

* Not specified

Other:

* No other concurrent lymphoma therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-10

CONTACTS AND LOCATIONS:
Overall Officials: Tillman Pearce, MD, Study Chair — Facet Biotech
Locations (1):
- Protein Design Labs, Inc., Freemont, California, United States